CLINICAL TRIAL: NCT03528824
Title: Randomised Controlled Trial on the Efficacy of Fenugreek Wraps in Symptomatic Primary Gonarthrosis
Brief Title: Fenugreek Wraps in Osteoarthritis of the Knee
Acronym: BoGon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Petra Klose, PhD, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BoGon
Record Dates: First submitted 2018-05-06; First posted 2018-05-18 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fenugreek wraps (Experimental): Daily application of fenugreek wraps for 1/2-2 hours per day, 4 weeks application
  Interventions: Other: Fenugreek wrap
- Diclofenac gel (Active Comparator): Daily application of diclofenac gel, 4 weeks application
  Interventions: Drug: Diclofenac Gel
- Usual care (No Intervention): no specific intervention

INTERVENTIONS:
Other: Fenugreek wrap — Daily application of fenugreek wraps for 1/2-2 hours per day, 4 weeks application
  Arms: Fenugreek wraps
Drug: Diclofenac Gel — Daily application of diclofenac gel, 4 weeks application
  Other Names: Diclofenac Emulgel
  Arms: Diclofenac gel

SUMMARY:
This randomised controlled trial aims to investigate the efficacy of fenugreek wraps in the treatment of primary symptomatic osteoarthritis of the knee. 81 patients will be randomised into one of 3 groups and apply fenugreek wraps or diclofenac gel daily for 4 weeks or receive only usual care. Efficacy will be measured using questionnaire on pain, disability,function, quality of life and pressure pain sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of the knee, Kellgren Lawrence stadium 2-3
* at least 50% of days with complaints in past 3 months
* initial pain intensity >45mm on a 100mm visual analoge scale

Exclusion Criteria:

* systemic medication with corticoids or immunosuppressive drugs
* systemic medication with chondroitinsulfate or glucosamine
* secondary arthrosis
* operation on the knee within the past 12 months
* injection within 4 weeks (cortisone) or 6 months prior (hyaluronic acid)
* severe comorbidities (tumor, psychiatric disorders etc.)
* participation in other studies, regarding gonarthrosis
* asthma
* pregnancy, breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  pain intensity measured on three 0-100mm visual analogous scales (actual, mean, worst pain)

SECONDARY OUTCOMES:
knee function (WOMAC) | 4 weeks
  physical everyday function using the validated WOMAC questionnaire
measure yourself medical outcome profile (MYMOP) | 4 weeks
  evaluation of symptoms and limitations
Quality of Life (SF-36) | 4 weeks
  health related quality of life with the validated SF-36 questionnaire
self-efficacy (ASES-D) | 4 weeks
  self-efficacy with the arthritis specific self efficacy scale in German
physical function (30second chair test) | 4 weeks
  validated test to measure how often patients can stand up from a chair in 30 seconds)
Course of Pain | 4 weeks
  measured by a diary including pain intensity on a visual analogue scale, medication
Pressure pain sensitivity | 4 weeks
  measured by an algometer at predefined areas
Adverse events Safety measure | 4 weeks
  safety measure
knee function (WOMAC) | 12 weeks
  physical everyday function using the validated WOMAC questionnaire
measure yourself medical outcome profile (MYMOP) | 12 weeks
  evaluation of symptoms and limitations
Quality of Life (SF-36) | 12 weeks
  health related quality of life with the validated SF-36 questionnaire
self-efficacy (ASES-D) | 12 weeks
  self-efficacy with the arthritis specific self efficacy scale in German
Course of Pain | 12 weeks
  measured by a diary including pain intensity on a visual analogue scale, medication
Adverse events | 12 weeks
  safety measure
Pain intensity | 12 weeks
  pain intensity measured on a three 0-100mmvisual analogous scales (actual, mean, worst pain)

CONTACTS AND LOCATIONS:
Locations (1):
- • Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine, University of Duisburg-Essen, Essen, Germany